CLINICAL TRIAL: NCT05052983
Title: A Double-Blind, Placebo-Controlled, Randomized Study to Assess the Durability of Effect and Safety of Nemolizumab for 24 Weeks in Subjects With Prurigo Nodularis
Brief Title: A Study to Evaluate the Durability of Response and Safety of Nemolizumab for 24 Weeks in Participants With Prurigo Nodularis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.203890; 2021-003928-32 (EudraCT Number)
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo Nodularis; Nemolizumab; CD14152
MeSH Terms: interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemolizumab (Experimental)
  Interventions: Drug: Nemolizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nemolizumab — Participants received either 1 [30 milligram (mg)] or 2 (2*30 mg) subcutaneous (SC) injection(s) of nemolizumab every 4 weeks (Q4W) for a period of 24 weeks (with last injection at Week 20). Participants received the same dosage (1 or 2 SC injections) as received in the lead-in LTE study RD.06.SPR.202699, as assigned by interactive response technology (IRT).
  Other Names: CD14152
  Arms: Nemolizumab
Drug: Placebo — Participants received either 1 (30 mg) or 2 (2*30 mg) SC injection(s) of placebo every 4 weeks for a period of 24 weeks (with last injection at Week 20). Participants received the same dosage (1 or 2 SC injections) as received in the lead-in LTE study RD.06.SPR.202699, as assigned by IRT.
  Arms: Placebo

SUMMARY:
The main objective of this study is to assess the long-term durability of response over a 24-week period following withdrawal of nemolizumab in participants with prurigo nodularis (PN) who previously responded to treatment in the Long-term-Extension (LTE) study RD.06.SPR.202699 (NCT05052983). The secondary objective of this study is to assess the safety of nemolizumab compared to placebo over a 24-week period in participants with PN who previously responded to treatment in the LTE study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who achieved a clinical response at Week 52 of the LTE study RD.06.SPR.202699, defined as:

   1. Investigator Global Assessment (IGA) score of 0 (clear) or 1 (almost clear) AND
   2. Greater than or equal to (>=)4-point improvement in weekly average of PP NRS score from baseline of the lead-in study Note: Lead-in study baseline is defined as baseline Peak Pruritus Numerical Rating Scale (PP NRS) score in the Phase 3 studies RD.06.SPR.202685 or RD.06.SPR.203065 for participants who rolled over into the LTE from these studies. For participants who entered the LTE study from the Phase 2 study RD.03.SPR.115828, the baseline PP NRS score at entry into the LTE study RD.06.SPR.202699 will be used
2. Participants with uninterrupted dosing of nemolizumab in the LTE study RD.06.SPR.202699 for 3 months before the Week 52 visit
3. Participants willing and able to transfer into the study at the time of completion of the Week 52 visit in the LTE study RD.06.SPR.202699
4. Female participants of childbearing potential (i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile) must agree to use an adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection. Adequate and approved methods of contraception applicable for the participant and/or her partner are defined in the Protocol
5. Female participants of non-childbearing potential must meet one of the following criteria:

   1. Absence of menstrual bleeding for 1 year prior to baseline without any other medical reason, confirmed with follicle-stimulating hormone (FSH) level in the postmenopausal range
   2. Documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least 3 months before the study
6. Participants willing and able to comply with all of the time commitments and procedural requirements of the clinical study protocol, including periodic weekly recordings by the participant using an electronic handheld device provided for this study.
7. Understand and sign an informed consent form (ICF) before any investigational procedure(s) are performed

Exclusion Criteria:

1. Participants who, during their participation in a prior nemolizumab study, experienced an adverse event which in the opinion of the Investigator could indicate that continued treatment with nemolizumab may present an unreasonable risk for the participant
2. Body weight less than (<) 30 kg (kilogram)
3. Receipt of prohibited medications, including rescue therapy, in the LTE study RD.06.SPR.202699 within 6 months of the Week 52 visit
4. Pregnant women (positive pregnancy test result at baseline visit), breastfeeding women, or women planning a pregnancy during the clinical study
5. Any medical or psychological condition that may put the participant at significant risk according to the Investigator's judgment, if he/she participates in the clinical study, or may interfere with study assessments (e.g., poor venous access or needle-phobia)
6. Planning or expected to have a major surgical procedure during the clinical study
7. Participants unwilling to refrain from using prohibited medications during the clinical study
8. History of alcohol or substance abuse within 6 months of baseline
9. Participants with confirmed or suspected COVID-19 infection within 2 weeks before baseline
10. Any condition the Investigator deems incompatible with participant participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Galderma Investigational Site 8521, Saint Joseph, Missouri, United States
- Austria (2):
  - Galderma Investigational Site 5471, Graz
  - Galderma Investigational Site 6158, Vienna
- France (3):
  - Galderma Investigational Site 5104, Brest
  - Galderma Investigational Site 5140, Nice
  - Galderma Investigational Site 6168, Valence
- Germany (3):
  - Galderma Investigational Site 5604, Berlin
  - Galderma Investigational Site 6082, Bonn
  - Galderma Investigational Site 6210, Heidelberg
- Poland (3):
  - Galderma Investigational Site 6052, Krakow
  - Galderma Investigational Site 6237, Ostrowiec Świętokrzyski
  - Galderma Investigational Site 5495, Rzeszów
- Galderma Investigational Site 6098, Ansan, South Korea
- Galderma Investigational Site 5069, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 14 study sites in 7 countries from 24 January 2022 to 11 September 2023.
Pre-assignment Details: A total of 34 participants from long-term extension (LTE) study RD.06.SPR.202699 (NCT05052983) were enrolled and treated in this study.
Groups:
- Nemolizumab: Participants received either 1 (30 milligram [mg]) or 2 (2*30 mg) subcutaneous (SC) injection(s) of nemolizumab every 4 weeks (Q4W) for a period of 24 weeks (with last injection at Week 20). Participants received the same dosage (1 or 2 SC injections) as received in the lead-in LTE study RD.06.SPR.202699 (NCT05052983), as assigned by interactive response technology (IRT).
- Placebo: Participants received either 1 (30 mg) or 2 (2*30 mg) SC injection(s) of placebo Q4W for a period of 24 weeks (with last injection at Week 20). Participants received the same dosage (1 or 2 SC injections) as received in the lead-in LTE study RD.06.SPR.202699 (NCT05052983), as assigned by IRT.
Period: Overall Study
Arm/Group | Nemolizumab | Placebo
Started | 18 | 16
Completed | 14 | 4
Not Completed | 4 | 12
Not completed — Lack of Efficacy | 3 | 12
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants.
Groups:
- Nemolizumab: Participants received either 1(30mg) or 2(2*30 mg) SC injection(s) of nemolizumab Q4W for a period of 24 weeks (with last injection at Week 20). Participants received the same dosage (1 or 2 SC injections) as received in the lead-in LTE study RD.06.SPR.202699 (NCT05052983), as assigned by IRT.
- Total: Total of all reporting groups
Arm/Group | Nemolizumab | Placebo | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (14.06) | 59.1 (13.41) | 59.5 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time From Baseline to Relapse Meeting At Least 1 of the Defined Criteria
Description: Time from baseline to relapse, defined as meeting at least 1 of the following criteria.
  1. Increase in (weekly average of the) PP NRS score >=4 points from baseline
  2. Increase in IGA score >=2 points from baseline. Time to relapse was censored at the last assessment of IGA and PP NRS prior to treatment discontinuation or use of prohibited medication
Time Frame: Baseline up to Week 24
Population: ITT population included all randomized participants. Here, "overall number of participants analyzed" signified participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 3 | 12
Days | NA [NA to NA] — Median, lower and upper limits of 95 percent (%) confidence interval (CI) could not be estimated due to insufficient data for time to relapse, as number of participants with relapse are only 3. | 112.50 [84.00 to 161.00]

2. Secondary Outcome: Percentage of Participants Maintaining Investigator Global Assessment (IGA) Success at Each Scheduled Visit
Description: IGA is a 5-point scale used by the investigator or trained designee to evaluate the global severity of PN. The Investigator reviewed the participant's skin and give a score of 0 (Clear), 1 (Almost clear), 2 (Mild), 3 (Moderate), or 4 (Severe). Treatment response/success was defined as 0 (clear) or 1 (almost clear).
Time Frame: Baseline up to Week 24
Population: ITT population included all randomized participants. Here, number analyzed signifies participants who were evaluable for given categories. Observed Cases (OC) analysis is applied here, where analysis is using all the observed data at each time point, no imputation for missing data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 18 | 16
Percentage of Participants
  At Week 4: number analyzed (Participants) | 17 | 15
  At Week 4 | 88.2 | 86.7
  At Week 8: number analyzed (Participants) | 17 | 16
  At Week 8 | 82.4 | 81.3
  At Week 12: number analyzed (Participants) | 17 | 15
  At Week 12 | 88.2 | 53.3
  At Week 16: number analyzed (Participants) | 16 | 11
  At Week 16 | 81.3 | 27.3
  At Week 20: number analyzed (Participants) | 15 | 7
  At Week 20 | 86.7 | 57.1
  At Week 24: number analyzed (Participants) | 14 | 5
  At Week 24 | 85.7 | 60.0

3. Secondary Outcome: Percentage of Participants With Increase in Peak Pruritus (PP) Numeric Rating Scale (NRS) Score of >= 4 Points From Baseline at Each Scheduled Visit
Description: Pruritus NRS is a scale that is used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a 11-point scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 18 | 16
Percentage of Participants
  At Week 4: number analyzed (Participants) | 13 | 13
  At Week 4 | 0 | 0
  At Week 8: number analyzed (Participants) | 13 | 14
  At Week 8 | 0 | 0
  At Week 12: number analyzed (Participants) | 16 | 12
  At Week 12 | 0 | 16.7
  At Week 16: number analyzed (Participants) | 15 | 12
  At Week 16 | 6.7 | 33.3
  At Week 20: number analyzed (Participants) | 14 | 6
  At Week 20 | 0 | 33.3
  At Week 24: number analyzed (Participants) | 10 | 5
  At Week 24 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to end of study (Week 32)
Description: The safety population included all randomized participants who receive at least 1 dose of study drug.
Arm/Group | Nemolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/16
Other Adverse Events (participants affected / at risk) | 11/18 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab (N=18) | Placebo (N=16)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab (N=18) | Placebo (N=16)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Administration site reaction (General disorders) | 1 | 0
Administration site erythema (General disorders) | 1 | 0
Injection site haematoma (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pustule (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Peak expiratory flow rate decreased (Investigations) | 0 | 1
Urinary lipids present (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 2 | 0
Diabetic macroangiopathy (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT05052983/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT05052983/SAP_001.pdf